CLINICAL TRIAL: NCT00814112
Title: GAGS - Glykosaminoglykaner Vid Sepsis
Brief Title: Glycosaminoglycans During Septic Shock - a Temporal Study
Acronym: GAGS
Status: Withdrawn | Type: Observational
Why Stopped: Lack of personell
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: GAGS 293/2008
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 septic shock: septic shock, ICU
- 2 controls: matched controls

SUMMARY:
We have previously shown that the plasma level of glycosaminoglycans (GAG) in septic shock patients are elevated compared to controls. The purpose of this study is to investigate the temporal dynamic of the blood level of GAG in ten septic shock patients. In addition, to assess the kinetics of GAG during septic shock we examine the liver function by galactose elimination capacity as well as excreted urinary GAG.

ELIGIBILITY:
Inclusion Criteria:

* 2 out of 4 SIRS criteria, where the circulatory criteria must be fulfilled
* Clinical sepsis is suspected
* Informed consent from relative
* Study subject must be over 18 years old

Exclusion Criteria:

* Pregnancy
* >24h post sepsis diagnosis
* Ongoing oral or intravenous cortisone treatment for more than one month.
* Malignancy with metastasis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Septic Shock
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11 (Estimated); Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Bodelsson, professor, Principal Investigator — Intensive Care Unit, Lund University Hospital, Sweden
Locations (1):
- Intensive Care Unit, Lund University Hospital, Lund, Sweden